CLINICAL TRIAL: NCT05572476
Title: Lurbinectedin Combined With Durvalumab in Pre-treated Patients With Extensive Stage Small-cell Lung Cancer
Acronym: LURBIMUNE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties, decline in the incidence of the studied pathology, active competitive clinical trials
Sponsor: Institut Bergonié (Other)
Collaborators: AstraZeneca (Industry); PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2022-01; 2022-001114-19 (EudraCT Number)
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer; Platinum-Sensitive Lung Small Cell Carcinoma; Extensive-stage Small-cell Lung Cancer
Keywords: small cell lung cancer; platinum sensitive
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; Etoposide

STUDY DESIGN:
Intervention Model Description: Randomized phase II study in which eligible patients will be randomized (2:1) according to two therapeutic strategies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A: treatment by lurbinectedin and durvalumab (Experimental): Patients with with platinum sensitive extensive stage small-cell lung cancer (SCLC) which failed one prior platinum-containing regimen will be treated by the association of lurbinectedin and durvalumab
  Interventions: Drug: Association of lurbinectedin and durvalumab
- Standard Arm B: treatment by carboplatin and etoposide (Other): Patients with with platinum sensitive extensive stage small-cell lung cancer (SCLC) which failed one prior platinum-containing regimen will be treated by the association of carboplatin and etoposide
  Interventions: Drug: Association of carboplatin and etoposide

INTERVENTIONS:
Drug: Association of lurbinectedin and durvalumab — A treatment cycles consists of 3 weeks (i.e. 21 days). Lurbinectedin will be administered by intravenous infusion on Day 1 every 3 weeks.
  Durvalumab will be administered by intravenous infusion on Day 1 every 3 weeks.
  Arms: Experimental Arm A: treatment by lurbinectedin and durvalumab
Drug: Association of carboplatin and etoposide — Treatment will be administered on a 21-days cycle basis up to a maximum of 6 cycles.
  Carboplatin will be administered by intravenous infusion on Day 1 every 3 weeks.
  Etoposide will be administered by intravenous infusion on Day 1-3 every 3 weeks
  Arms: Standard Arm B: treatment by carboplatin and etoposide

SUMMARY:
Multicenter, prospective, open-labeled, 2-arm, randomized non-comparative (2:1) phase II trial assessing the efficacy of lurbinectedin in association with durvalumab

DETAILED DESCRIPTION:
Multicenter, prospective, open-labeled, 2-arm, randomized non-comparative (2:1) phase II trial assessing the efficacy of lurbinectedin in association with durvalumab in pre-treated patients with platinum sensitive extensive stage small-cell lung cancer (SCLC) which failed one prior platinum-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histology: confirmed diagnosis of extensive stage SCLC which failed one prior platinum-containing regimen,
2. Recurrent and platinum-sensitive SCLC: defined as those patients with SCLC recurrence at least 90 days from the last dose of platinum-based chemotherapy. Definition of platinum-sensitive disease is patient with at least 90 days of progression-free duration after finishing first-line platinum-based chemotherapy
3. Patients must have received as first line a combo with platinum+ etoposide + PD_L1 inhibitor
4. Metastatic or unresectable locally advanced disease, not ammenable to curative therapy,
5. Age ≥ 18 years,
6. Eastern Cooperative Oncology Group ≤ 1,
7. Life expectancy > 3 months,
8. Patients must have measurable disease as per RECIST v1.1.
9. Documented disease progression according to RECIST v1.1 before study entry,
10. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment for neoplastic disease and/or radiotherapy,
11. Adequate hematological, renal, metabolic and hepatic function
12. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. Both women and men must agree to use a highly effective method of contraception ,
13. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, concomitant endometrial carcinoma stage IA grade 1, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
14. Recovery to grade ≤ 1 from any adverse event derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the NCI-CTCAE, version 5,
15. Body weight >30kg
16. Voluntarily signed and dated written informed consent prior to any study specific procedure,
17. Patients with a social security in compliance with the French law.

Exclusion Criteria:

1. Previous treatment with lurbinectedin,
2. Current or prior use of immunosuppressive medication including any use of oral glucocorticoids, within 14 days before the first dose of durvalumab,
3. Active or prior documented inflammatory bowel disease,
4. Has an active autoimmune disease requiring systemic treatment within the past 2 years,
5. Has evidence of active non-infectious pneumonitis,
6. Has an active or ongoing infection requiring systemic therapy,
7. Currently active bacterial or fungus infection, HIV1, HIV2, hepatitis A or hepatitis B or hepatitis C infections,
8. Symptomatic untreated, or steroid-requiring, or progressing central nervous system malignancy is excluded.
9. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding,
10. Previous enrolment in the present study,
11. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
12. Has received a live vaccine within 30 days prior to the first dose of trial treatment,
13. Known hypersensitivity to any involved study drug or any of its formulation components,
14. Tumors not accessible for biopsy,
15. Active infection including tuberculosis,
16. Person under judicial protection or deprived of liberty,
17. Concomitant use of strong inhibitors or inductors of cytochrome CYP3A4 taken within 21 days prior to the first dose of study drug,
18. Uncontrolled symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, myocardial infarction, clinically significant valvular heart disease,
19. Intermittent or continuous oxygen requirement,
20. Presence of any external drainage,
21. Known myopathy,
22. Concomitant administration of any other antineoplastic therapy, other investigational agents, immunosuppressive therapies, Aprepitan or any other NK-1 antagonist,
23. Major surgical procedure within 28 days prior to the first dose of durvalumab.
24. History of allogenic organ transplantation,
25. History of leptomeningeal carcinomatosis,
26. QT interval corrected for heart rate using Fridericia's formula ≥470 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of lurbinectedin combined with durvalumab | 6 months
  Antitumor activity will be assessed in terms of of 6-month progression-free rate (rate of complete or partial responses or stable disease more than 24 weeks, as per RECIST v1.1 criteria) after blinded centralized radiological review

SECONDARY OUTCOMES:
6-months objective response for experimental Arm | 6 months
  Objective response is defined as the proportion of patients with complete response (CR) or partial response (PR) observed at 6 months, based on RECIST 1.1 criteria.
Best overall response for experimental Arm | Throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best response across all time points (RECIST 1.1). The best overall response is determined once all the data for the patient is known (RECIST 1.1).
1-year progression-free survival for experimental Arm | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
2-year progression-free survival for experimental Arm | 2 years
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
1-year overall survival for experimental Arm | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
2-years overall survival for experimental Arm | 2 years
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
Safety profile for experimental Arm: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5.
Safety profile for standard Arm: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5.
Assessment of the antitumor activity of carboplatin combined with etoposide | 6 months
  Antitumor activity will be assessed in terms of of 6-month progression-free rate (rate of complete or partial responses or stable disease more than 24 weeks, as per RECIST v1.1 criteria) after blinded centralized radiological review
6-months objective response for standard Arm | 6 months
  Objective response is defined as the proportion of patients with complete response (CR) or partial response (PR) observed at 6 months, based on RECIST 1.1 criteria.
Best overall response for standard Arm | Throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best response across all time points (RECIST 1.1). The best overall response is determined once all the data for the patient is known (RECIST 1.1).
1-year progression-free survival for standard Arm | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
2-year progression-free survival for standard Arm | 2 years
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
1-year overall survival for standard Arm | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
2-years overall survival for standard Arm | 2 years
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
Tumor immune cells levels | before treatment onset, at cycle 2 days 1, cycle 3 day 1 and at progression (each cycle is 21 days)
  Levels of immune cells in tumor will be measured by immunohistochemistry
Blood cytokines levels | before treatment onset, at cycle 2 days 1, cycle 3 day 1 and at progression (each cycle is 21 days)
  Levels of cytokines in blood will be measured by ELISA
Blood lymphocytes levels | before treatment onset, at cycle 2 days 1, cycle 3 day 1 and at progression (each cycle is 21 days)
  Levels of lymphocytes in blood will be measured by flow cytometry
Blood kynurenine levels | before treatment onset, at cycle 2 days 1, cycle 3 day 1 and at progression (each cycle is 21 days)
  Levels of kynurenine in blood will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France